CLINICAL TRIAL: NCT05662072
Title: Effects of Motor Imagery and Action Observation on Respiratory Parameters
Brief Title: Motor Imagery and Action Observation in Respiratory Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Luis Suso, Principal investigator, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2022-12-05; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Respiratory Function; Motor Imagery; Action Observation Training
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motor imagery (Experimental): Motor imagery of inspiratory and expiratory exercises, 10 series of 1 minute.
  Interventions: Behavioral: Motor imagery
- Action observation (Experimental): Action observation of inspiratory and expiratory exercises, 10 series of 1 minute.
  Interventions: Behavioral: Action observation
- Placebo Observation (Placebo Comparator): Placebo visualization of nature video, 10 minutes.
  Interventions: Other: Placebo Intervention

INTERVENTIONS:
Behavioral: Motor imagery — Mental imagery of respiratory exercises
  Arms: Motor imagery
Behavioral: Action observation — Action observation of respiratory exercises
  Arms: Action observation
Other: Placebo Intervention — Placebo observation
  Arms: Placebo Observation

SUMMARY:
The principal aim of this study was to asses the effects of motor imagery and action observation training on ventilatory and functional capacity through a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60
* Healthy and with no respiratory pathology subjects

Exclusion Criteria:

* Any cognitive impairment that hindered viewing of audiovisual material.
* Difficulty understanding or communicating.
* Presence of systemic pathology, Central Nervous System or rheumatic disease.
* Inadequate understanding of the Spanish language to follow instructions for measuring and treatment.
* Collaboration of pregnant women.
* Underage subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-05 (Estimated); Primary Completion 2023-02-04 (Estimated); Study Completion 2023-03-05 (Estimated)

PRIMARY OUTCOMES:
Change from Forced vital capacity physiological parameter | Preintervention and postintervention (after the 10 minutes intervention)
  With spirometry
Change from FEV1 physiological parameter | Preintervention and postintervention (after the 10 minutes intervention)
  With spirometry